CLINICAL TRIAL: NCT04139980
Title: Virtual Reality Device for Rehabilitation of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chen Lin, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300003889
Record Dates: First submitted 2019-10-02; First posted 2019-10-25 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality supported therapy (Experimental): The Virtual Reality (VR) interface will be used during patients stay at the rehabilitation center. A research employee will install the VR system in the patient's room. Participants will be comfortable sitting while in VR session. Each interface consists of a head mounted display (HMD) allowing participants to see their arms and legs represented in the virtual environment. Participants will be able to control their virtual legs using hand controllers, which will allow them to "walk" through several virtual environments and gather "points" (no additional gaming elements are included).
  Interventions: Other: Virtual Reality (VR)

INTERVENTIONS:
Other: Virtual Reality (VR) — Each VR session is 30 minutes long. Participants are able to pause or discontinue at any time. Each participant will receive one VR sessions five times per week over the course of a two-week period.
  Other Names: HTC Vive VR System

SUMMARY:
This study will evaluate the potential efficacy and safety of using virtual reality gaming in conjunction to standard therapy regimen care as an approach to promote upper-limb motor recovery, cognitive function and quality of life after stroke. The investigators believe that allowing users to interact with a computer-simulated reality environment will result in a pleasant experience, which will likely result in motivation and therapy engagement.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to the UAB Hospital, older than 18 years old, with a diagnosis of stroke
* Patient with unilateral upper extremity weakness
* Patients that after evaluation by Physical and Occupational professionals were admitted to rehabilitation facility "Spain Rehabilitation Center".

Exclusion Criteria:

* Patients with severe cognitive impairment
* Patient with orthopedic impairment (i.e. marked arthritis)
* Patient with visual disorders limiting therapy session
* Those for whom voluntary arm movement would cause sufficient discomfort (>4/10) that could prevent trial completion will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Change in Upper-limb and hand motor function | Change from NIHSS measured at baseline visit, one week after final VR session, and three months following discharge. Totals are summed to determine the range:0= No stroke, 1-4 = Minor, 5-15 = Moderate, 15-20= Moderate to Severe; and 21-42 = Severe
  National Institutes of Health Stroke Scale (NIHSS)
Change in upper-limb and hand motor function | Change from motricity index measured at baseline visit, one week following final VR session, and three months following discharge from rehabilitation center
  Motricity Index
Change in upper-limb and hand motor function | Change from Action Research Arm Test measured at baseline visit, one week following final VR session, and three months following discharge from rehabilitation center
  Action Research Arm Test
Change in upper-limb and hand motor function | Change from Nine hole Peg test measured at baseline visit, one week following final VR session, and three months following discharge from rehabilitation center
  Nine hole Peg test
Change in upper-limb and hand motor function | Change from Fugl-Meyer Assessment measured at baseline visit, one week following final VR session, and three months following discharge from rehabilitation center
  Fugl-Meyer Assessment
Change in upper-limb and hand motor function | Change from m-RS measured at baseline, one wee following final VR session, and three months following discharge. The score is based on symptoms with a 0 provided for no symptoms up to a 5 provided for severe disability; bedridden, requires constant care.
  Modified Rankin Scale (m-RS)

SECONDARY OUTCOMES:
Change in cognitive function | Change from MOCA measured at baseline, one week following final VR session, and three months following discharge. The scores are summed. The range is: 27-30=Normal; 18-26=Mild impairment; 10-17=Moderate impairment; <10=Severe
  Montreal Cognitive Assessment (MOCA)
Change in activities of daily living (ADL) and quality of life | Change in SIS measured at baseline, one week after final VR session, and three months after discharge. Range is 0-100. Higher scores indicate better ADL and quality of life. Formula: Actual raw score - lowest possible score/Possible raw score)*100
  Stroke Impact Scale (SIS)
Change in depression | Change from PHQ9 measured at baseline, one week following final VR session, and three months following discharge. Scores are totaled with higher score being severe. 5-9 = Mild, 10-14 = Moderate, 15-19 = Moderately severe, 20-27 = Severe
  Patient Health Questionnaire 9 (PHQ9)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Lin, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Spain Rehabilitation Center, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided